CLINICAL TRIAL: NCT02794493
Title: A Phase III Randomized, Placebo-controlled, Double-blind Trial to Determine the Effectiveness of Traditional Chinese Medicine Formula LC09 for Treatment of Capecitabine-Induced Hand and Foot Syndrome
Brief Title: Treatment of Hand and Foot Syndrome With Traditional Chinese Medicine Formula LC09 in Patients Who Are Receiving Capecitabine for Colorectal and/or Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Yanni Lou, Attending Doctor, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015BAI04B07
Record Dates: First submitted 2016-05-26; First posted 2016-06-09 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Hand Foot Syndrome
MeSH Terms: conditions — Hand-Foot Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Arm I (Experimental): Patients receive Traditional Chinese Medicine Formula LC09 by soaking their affected hand and feet 20 min twice daily.
  Interventions: Drug: Traditional Chinese Medicine Formula LC09
- Arm II (Placebo Comparator): Patients receive placebo by soaking their affected hand and feet 20 min twice daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Traditional Chinese Medicine Formula LC09
  Arms: Arm I
Other: Placebo
  Arms: Arm II

SUMMARY:
RATIONALE: Hand foot syndrome may be treated or reduced by soaking Traditional Chinese Medicine Formula LC09 in patients receiving capecitabine for colorectal and/or breast cancer.

PURPOSE: This randomized phase III trial is studying soaking Traditional Chinese Medicine Formula LC09 to see how well they work compared to placebos in preventing hand-foot syndrome in patients who are receiving capecitabine for colorectal or breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

OBJECTIVES: Determine whether Traditional Chinese Medicine Formula LC09 can treat or reduce the severity of capecitabine-caused hand foot syndrome.

Evaluate the potential toxicity of Traditional Chinese Medicine Formula LC09. OUTLINE: This is a multicenter, randomized, double-blind, placebo-controlled study. Patients are randomized to 2 treatment arms.

Arm I: Patients receive Traditional Chinese Medicine Formula LC09 by soaking their affected hand and feet 20 min twice daily.

Arm II: Patients receive placebo by soaking their affected hand and feet 20 min twice daily.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following criteria to be eligible for the study:

1. Histologically confirmed colorectal cancer or breast cancer, of which colorecta cancer is advanced or undergoing adjuvant therapy after radical resection and breast cancer is at the stage of recurrence or metastasis;
2. Level 1 or above HFS after receiving capecitabine as part of routine standard care;
3. Plan to receive capecitabine as part of routine more than 2 weeks;
4. ECOG performance status 0-2;
5. Life expectancy greater than or equal to 3 months;
6. No serious heart, liver, kidney and other important viscera dysfunction, as defined below:

   * absolute neutrophil count greater than or equal to 1.5 x 10(9)/L
   * platelet count greater than or equal to 100 x 10(9)/L
   * hemoglobin greater than or equal to 9.0 g/dL
   * total bilirubin less than or equal to 1.5 times the ULN
   * AST/SGOT and ALT/SGPT less than or equal to 2.5 times the ULN (or less than or equal to 5 times the ULN if liver function abnormalities due to underlying malignancy)
   * creatinine less than or equal to 1.5 times the ULN
   * creatinine clearance greater than or equal to 60 ml/min (by Cockcroft-Gault)
7. Ability to cooperate with HFS grade evaluation, understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Subjects meeting any of the following criteria are ineligible for study entry:

1. Concurrent with level 1 or above peripheral neuropathy (such as diabetic neuropathy or chemotherapy induced peripheral neuropathy);
2. Other acute or chronic inflammatory conditions or infections of the hands or feet that would complicate safety, application of topical creams, or study endpoints;
3. Currently taking other treatment for PPE (including topical urea cream, pyridoxine, celecoxib, compound matrine injection and deproteinized calf blood extractive injection);
4. History of severe or uncontrolled organic disease or infection, such as heart, pulmonary or renal failure that cause the termination of chemotherapy;
5. Pregnant (positive pregnancy test) or nursing women;
6. Participating in other clinical trial currently or within 4 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
Grade of hand foot syndrome over time as measured by NCI CTCAE version 4.03 PPE syndrome criteria | Once daily until the date that the consecutive 2 cycles of capecitabine-containing chemotherapy ended (up to 6 weeks)
  Grading of PPE by NCI CTC criteria is collected on a diary card that subjects fill out once daily. Investigators assess and fill the grading into the case report form every week.
Assessment of patient reported pain using a 1-10 score. | Once daily until the date that the consecutive 2 cycles of capecitabine-containing chemotherapy ended(up to 6 weeks)
  Assessment of patient reported pain using a 1-10 score is collected on a diary card that subjects fill out once daily.

SECONDARY OUTCOMES:
Instrumental Activities of Daily Living Scale | Baseline and after the intervention completed (up to 6 weeks)
  Performance assessment on 8 daily tasks
Dermatology Life Quality Index (DLQI) Total Score | Baseline and after the intervention completed (up to 6 weeks)
  The DLQI is a 10-item general dermatology questionnaire that assess health related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). The DLQI item response options are rated by the participant from 0 (not at all/not relevant) to 3 (very much) with a total score range of 0 (best) to 30 (worst); higher scores indicate poor quality of life.
Chemotherapy completion rate | After the intervention completed (up to 6 weeks)
  Proportion of patients having tolerated established 2-week chemotherapy in each arms.
Incidence of reduced dosage of capecitabine thereby | After the intervention completed (up to 6 weeks)
  Reduced dosage of capecitabine thereby because of hand foot syndrome
Incidence of cessation of capecitabine thereby | After the intervention completed (up to 6 weeks)
  Cessation of capecitabine thereby because of hand foot syndrome

REFERENCES:
- [Derived] Yu R, Wu X, Jia L, Lou Y. Effect of Chinese Herbal Compound LC09 on Patients With Capecitabine-Associated Hand-Foot Syndrome: A Randomized, Double-Blind, and Parallel-Controlled Trial. Integr Cancer Ther. 2020 Jan-Dec;19:1534735420928466. doi: 10.1177/1534735420928466. PMID 32597691